CLINICAL TRIAL: NCT03770442
Title: Effect of Early Rehabilitation Using an Active/Passive Cycling Device on Muscle Wasting in the Critically Ill: A Randomised Controlled Study
Brief Title: Muscle Wasting in the Critically Ill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Ingeborg Welters, Senior Lecturer, Institute of Aging and Chronic Disease, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UoL001367
Record Dates: First submitted 2018-10-15; First posted 2018-12-10 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Muscle Weakness
Keywords: ICU acquired weakness (ICU-AW); FES; Functional Electrical Stimulation; Rehabilitation
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Ultrasound images will be labelled by their participant number, and not by intervention. Therefore, when image analysis takes place, the investigators will not know whether the images come from somebody who received cycling sessions or the control group.
  Tissue samples will be treated in the same way.
  In follow up sessions, participants will be asked not to reveal if they can remember whether they cycled or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cycling with FES (Experimental): Ten sessions of 14 days in patients consented within 48 hours of arriving in critical care who are sedated and mechanically ventilated with a diagnosis of sepsis from any source.
  Sessions last a maximum of 30 minutes (with an ideal minimum of 20 minutes), using the Restorative Therapies (RT) 300 Supine with the Sage 12-channel stimulator. Stimulation will provided to the quadriceps, hamstrings, calves and abdomen. Both legs and both sides of the abdomen will be stimulated. Stimulation current settings are individualised for each patient and each muscle group.
  These patients will also receive their routine physiotherapy that they would have received if they were in the control group (or not in the trial at all).
  Interventions: Device: Cycling with FES
- Control - routine physiotherapy (Active Comparator): Usual daily physiotherapy, consisting of limb care and mobilisation, and respiratory care and exercises as appropriate.
  Interventions: Other: Routine physiotherapy

INTERVENTIONS:
Device: Cycling with FES — As described already
  Other Names: RT-300 Supine; Restorative Therapies
  Arms: Cycling with FES
Other: Routine physiotherapy — As described already
  Arms: Control - routine physiotherapy

SUMMARY:
Muscle wasting is a common consequence of critical illness, and has a profound impact upon the rehabilitation of those who survive admission to critical to care. The investigators intend to assess if the application of 10 sessions over two weeks of passive cycling with electrical stimulation to the lower limbs and abdomen can prevent muscle loss, or at least cause less muscle loss, compared to patients who receive standard daily sessions of physiotherapy. This will be done by comparing the changes in muscle size on ultrasound between the two groups, comparing functional measures at a 3 month follow up, and by performing translational research using tissue samples taken during the study.

DETAILED DESCRIPTION:
Patients are mechanically ventilated and sedated with a diagnosis of sepsis (from any source) will be eligible for this study. Provided they meet the inclusion criteria, they will be randomised within 48 hours of admission, to either ten 30 minute sessions of passive cycling with functional electrical stimulation (FES) to the thighs, hamstrings, calves and abdomen over a 14 day period, or to a control group of routine physiotherapy. The trial group will also receive this physiotherapy.

On admission to the study, all patients will receive on day 1:

Ultrasound measurements of:

Rectus femoris cross-sectional area Thickness of rectus femoris and vastus intermedius Thickness, pennation angle and derived fascicle length of vastus lateralis and medial head of gastrocnemius Thickness of rectus abdominis. Thickness of diaphragm

A blood sample taken from an arterial line A urine sample taken from a urinary catheter A muscle biopsy taken from the right vastus lateralis

They will then receive ten 30 minute sessions of passive cycling with functional electrical stimulation over 14 days, or a control group will receive routine physiotherapy during this period.

Repeat ultrasounds will be taken at days 3, 5, 7, 10 and 14. Repeat blood and urine sampling at days 5, 10 and 14. Repeat muscle biopsy at day 14.

All cycling, ultrasounds and tissue sampling will end on day 14 regardless of the ventilator status of the patient.

In patients who survive to be discharged from critical care, they will be followed up at 3 months for:

Repeat ultrasound scan of all muscles listed Six minute walk test Hand grip and lower limb dynamometry, Balance testing (by standing upright on a pressure plate for 20 seconds) Psychological assessment using the 36 item Short Form (SF-36) questionnaire

Tissue sampling will be stored in the University of Liverpool for analysis of biomarkers of muscle damage and loss between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited in the Intensive Care Unit of the Royal Liverpool University Hospital. All patients will be over 18, and have a critical illness that requires mechanical ventilation with an initial period of sedation. This study will focus on patients with a definite or suspected case of sepsis from any source.

Sepsis has been recently redefined as: "Life threatening organ-dysfunction caused by dysregulated host response to infection" whilst septic shock has become a subset of sepsis, defined as: "circulatory and cellular/metabolic dysfunction associated with a higher risk of mortality(44).

For the purposes of this study, a patient will be regarded as septic if they have evidence of infection-related organ failure (e.g. sepsis-associated coagulopathy, altered mental state, cardiovascular dysfunction, acute kidney injury, and altered liver function) and require invasive mechanical ventilation with either definite or suspected evidence of infection. This is to allow prompt treatment with FES rather than waiting for a positive microbiological result to be obtained.

Within the definition of sepsis "from any source" a list of following is illustrative but not exhaustive:

* Urogenital sepsis (including urosepsis, pyelonephritis, endometritis and chorioamnionitis)
* Pneumonia (including community acquired, hospital acquired, and aspiration pneumonia. Ventilator associated pneumonia would be excluded.)
* Neurological infections such as encephalitis and meningitis.
* Cellulitis, osteomyelitis and infections of soft tissue NOT affecting the lower limb.
* Surgical infections, including post-operative laparotomy with evidence of peritoneal soiling, and evidence of infection prior to the operation, in patients who require 2 or more organ system support after the operation.
* Intra-abdominal sepsis, including biliary sepsis, hepatitis, and acute pancreatitis. In the case of acute pancreatitis, evidence of infection is required to fulfil the criteria. Acute pancreatitis with sterile tissue/fluid samples would not be suitable.

Exclusion Criteria:

* Patients under 18
* Patients who decline consent
* Pregnancy
* Neuromuscular disease
* Rhabdomyolysis
* Lower limb trauma
* Patients unlikely to survive to 96 hours post admission
* Consent unobtainable within 48 hours of admission
* Morbid obesity (BMI>40).
* Presence of a pacemaker or Implantable Cardiac Defibrillator (ICD).
* Unlikely to be mechanically ventilated for more than 48 hours.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound assessment of rectus femoris - Change in cross sectional area (cm2) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Measurement of cross-sectional area of rectus femoris (cm2)
Ultrasound assessment of rectus femoris - Change in muscle layer thickness (cm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Measurement on muscle layer thickness of rectus femoris (cm)
Ultrasound assessment of anterior thigh musculature - Change in muscle layer thickness (cm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Measurement of combined muscle layer thickness of rectus femoris and vastus intermedius (cm)
Ultrasound assessment of vastus lateralis - change in muscle layer thickness (cm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Measurement of the thickness of the vastus lateralis between the superficial and deep aponeuroses (cm)
Ultrasound assessment of vastus lateralis - change in fascicle pennation angle (degrees) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Measurement of the pennation angle of the muscle fascicles as they insert into the deep aponeuroses of the vastus lateralis muscle (degrees)
Ultrasound assessment of vastus lateralis - change in fascicle length (cm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  This is a single measure, derived by trigonometry (the Sine of the pennation angle multiplied by the muscle thickness).
Ultrasound assessment of the medial head of gastrocnemius - change in muscle thickness (cm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Measurement of the thickness of the medial head of the gastrocnemius between the superficial and deep aponeuroses (cm)
Ultrasound assessment of the medial head of gastrocnemius - change in fascicle pennation angle (degrees) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Measurement of the pennation angle of the muscle fascicles as they insert into the deep aponeuroses of the medial head of gastrocnemius (angles)
Ultrasound assessment of the medial head of gastrocnemius - change in fascicle length (cm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  This is single measure which is mathematically derived by trigonometry using the known pennation angle (degrees) and thickness (cm): the Sine of the pennation angle multiplied by the muscle thickness.
Ultrasound assessment of the rectus abdominis muscle - change in muscle layer thickness (cm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Measurement of rectus abdominis muscle layer thickness - (cm)
Diaphragm thickness assessment by ultrasound - change in end expiratory thickness (mm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Assessment of thickness at end expiration (mm)
Diaphragm thickness assessment by ultrasound - change in end inspiratory thickness (mm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Assessment of thickness at end inspiration (mm)
Diaphragm thickness assessment by ultrasound - change in thickening fraction (%) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Assessment of thickening fraction, derived mathematically from thicknesses at inspiration and expiration (%)
Ultrasound assessment of change in diaphragmatic excursion (cm) | Ultrasounds taken on day 1, 3, 5, 7, 10 and 14, and at 3 month follow up.
  Assessment of maximal excursion of diaphragm, measured with M-mode ultrasonography (mm)

SECONDARY OUTCOMES:
Measurement of change in blood biomarkers (microRNA analysis for markers of muscle loss, expressed as a percentage fold increase/decrease compared to baseline). | Samples taken on days 1, 5, 10 and 14
  Blood samples taken during the study period and analysed for markers of muscle loss/degradation
Measurement of change in urinary biomarkers (microRNA analysis for markers of muscle loss, expressed as a percentage-fold increase/decrease compared to baseline). | Samples taken on days 1, 5, 10 and 14
  Blood and urine samples taken during the study period and analysed for markers of muscle loss/degradation
Measurement of the number of biomarkers expressed from muscle biopsies (microRNA analysis for markers of muscle loss, expressed as the number and type of micro-RNAs expressed within the samples). | Samples taken on day 1 and 14
  Muscle biopsy samples taken during the study period and analysed for markers of muscle loss/degradation. Number and type of micro-RNAs to be noted).
Measurement of muscle fibre cross sectional area from muscle biopsies (mm2) | Samples taken on day 1 and 14
  Histological staining and analysis of muscle fibre composition, expressed in square millimetres and as a percentage-fold increase/decrease compared to baseline).
Follow up testing - Distance achieved in a 6 minute walk test, metres) | At 3 month follow up
  Distance achieved during a 6 minute shuttle walk of 20 metres length
Follow up testing - Hand grip dynamometry (hand grip strength, Newtons) | At 3 month follow up
  Strength of hand grip in both hands
Follow up - Lower limb strength assessment - Force generated at maximal contraction for knee extension (Newtons) | At 3 month follow up
  Strength of extension at the knee in both legs using a hand held dynamometry device (microFET 2 wireless device). Measured in Newtons.
Follow up testing - Balance assessment - Comparison of changes in center of pressure on a pressure plate. | At 3 month follow up
  Comparison of changes in centre of pressure on a pressure plate. The centre of pressure is measured over 20 seconds with the participant standing still. Maximal variation in lateral and anterior-posterior sway is recorded by the pressure plate.
Follow up testing - Psychological assessment - Comparison of total scores obtained from the SF-36 questionnaire (maximum score 100, minimum score zero). | At 3 month follow up
  Comparison of scores obtained from the SF-36 questionnaire between the two groups. A lower score indicates greater disability.
Follow Up - Maximal Inspiratory Pressure monitoring in kilopascals (kPa) | At 3 month follow up
  Using the Power Breathe K2 device
Incidence of delirium during the trial period - using the CAM-ICU tool. | Days 1-14
  Assessed by twice daily Cambridge Assessment Method for the ICU (CAM-ICU) assessments
Incidence of renal replacement therapy during the trial period | Days 1-14
  Daily monitoring to see if patient has required renal replacement therapy (defined as either haemofiltration or haemodialysis).
Total dose of noradrenaline given per day | Day 1-14
  Daily monitoring of doses of inotropic and vasopressor drugs
Overall fluid balance (in mls) at the end of each study day | Day 1-14
  Daily noting of 24 hour fluid balance
Total Insulin doses (in international units) required per day | Day 1-14
  Daily monitoring of exogenous insulin requirements
Blood glucose concentration (mmol/L) | Day 1-14
  Daily monitoring of glucose levels
Heart rate variability | Days 1 - 14 but only on the days where cycling takes place (ten sessions)
  Measured via a wireless skin patch
Safety - number of times an endotracheal/tracheostomy tube is dislodged during the cycling sessions | Days 1 - 14 but only on the days where cycling takes place (ten sessions)
  Expressed as a simple count of how many times an airway device dislodges
Safety - number of times an nasogastric tube is dislodged during the cycling sessions | Days 1 - 14 but only on the days where cycling takes place (ten sessions).
  Expressed as a simple count of how many times a nasogastric feed tube dislodges.
Safety - number of times an a central or arterial line device is dislodged during the cycling sessions | Days 1 - 14 but only on the days where cycling takes place (ten sessions).
  Expressed as a simple count of how many times a central or arterial line dislodges.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg D Welters, Principal Investigator — University of Liverpool
Locations (1):
- Intensive Care Unit, Royal Liverpool University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Translational research will take place in the Institute of Aging and Chronic Disease. Only the participant number of the sample will be shared with any staff working with tissue samples.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT03770442/Prot_SAP_000.pdf